CLINICAL TRIAL: NCT04770337
Title: STARSTIM: SAFETY AND THERAPEUTIC MEASURES OF TRANSCRANIAL CATHODAL DIRECT CURRENT STIMULATION (TDCS) IN PATIENTS WITH REFRACTORY FOCAL EPILEPSY
Brief Title: Pivotal-Safety and Therapeutic Measures of tDCS in Patients With Refractory Focal Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroelectrics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE001
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Refractory Epilepsy; Focal Seizure; Seizures, Focal; Seizures; Epilepsy in Children; Epilepsy; Epilepsy, Tonic-Clonic
Keywords: Epilepsy; Focal seizure; Seizure
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures; Epilepsy; Epilepsy, Tonic-Clonic

STUDY DESIGN:
Intervention Model Description: multiple site, randomized, double blinded parallel-group controlled study
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized in a 1:1 ratio to receive an active STARSTIM treatment or a sham treatment. Neither the study investigator nor subject shall be notified of the treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sham treatment (Sham Comparator): Subjects will be randomized in a 1:1 ratio to receive an active STARSTIM treatment or a sham treatment.
  Interventions: Device: Sham Device
- STARSTIM device treatment (Experimental): Subjects will be randomized in a 1:1 ratio to receive an active STARSTIM treatment or a sham treatment.
  Interventions: Device: STARSTIM device

INTERVENTIONS:
Device: STARSTIM device — Cathodal Transcranial Direct Current Stimulation (tDCS). Transcranial direct current stimulation (tDCS) is a form of neurostimulation which uses constant, low current delivered to the brain area of interest via electrodes on the scalp.
  Arms: STARSTIM device treatment
Device: Sham Device — Intervention which uses enough currents to generate a sensory feedback similar to that of active stimulation via electrodes on the scalp
  Arms: Sham treatment

SUMMARY:
This is a multiple site, randomized, double blinded parallel-group controlled study. The purpose of this study is to evaluate efficacy, safety, and tolerability of repeated, daily sessions with the STARSTIM device, which delivers transcranial cathodal direct current stimulation (tDCS). Subjects will be treated with STARTSTIM or sham device for 10 sessions over a 2-week period. The subjects will be followed for an additional 10 weeks post treatment. Quality of Life questionnaires and adverse events will be collected and evaluated.

DETAILED DESCRIPTION:
Study design is an evaluation of the STARSTIM device (tDCS) in subjects over 9 years of age, diagnosed with epilepsy with focal seizures with or without focal to bilateral tonic clonic seizures. Seizure diaries will be collected for 12 weeks to establish a rate of seizure for each subject prior to treatment. Subjects will be randomized in a 1:1 ratio to receive an active STARSTIM treatment or a sham treatment. Neither the study investigator nor subject shall be notified of the treatment assignment. Treatment will be done daily at the investigator's site for 10 days. A Seizure Diary will be maintained through the course of the treatment and the follow up period. Subjects will have 3 follow up visits to evaluate their seizure rate, adverse events, medications and quality of life. A Data Safety Monitoring Board will be utilized to evaluate safety events through study milestones. Seizure frequency rates pre, during and post treatment will be evaluated for both the active and sham treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. 9 years old or older
2. Diagnosis of epilepsy with focal seizures with or without focal to bilateral tonic clonic seizures (International League Against Epilepsy classification). Diagnosis established by both clinical history and an EEG consistent with focal seizures.

   Note: A normal interictal EEG is consistent with focal seizures, if other data is adequate to provide localization.
3. Epilepsy is refractory to treatment, defined as: failure to achieve adequate seizure control despite demonstrated compliance, according to medical records, on at least two (2) FDA-approved ASDs at a daily dose considered therapeutic for the patient's demographic according to package labeling, within approximately the last 3 years.
4. Seizure frequency ≥3 per month, over the past year.
5. Currently on ≥1 ASDs with no changes in antiepileptic drug doses in the 3 weeks prior to baseline visit in the study and no planned dose changes during the trial. Changes after baseline visit are permitted only if clinically necessary.
6. An MRI scan of the brain using 1.5 Tesla magnet, or greater, with T1, T2, and FLAIR sequences, performed within past 3 years and more recently than any craniotomy or skull burr hole procedure.
7. Seizure focus that allows design of an appropriate stimulation montage. Note: Seizure focus can be identified within a lobe, or 2 adjacent lobes. Identification of the border of the seizure focus can be approximate (+/- 2 gyri).
8. Available seizure history and supporting data
9. All female study subjects of child-bearing age are required to have a pregnancy test. Additionally, all females of childbearing potential will be required to use an effective method of birth control (defined as having a documented failure rate of <=1%; for women using enzyme-inducing ASDs hormonal contraceptives will not be considered as effective).
10. Written informed consent obtained from study subject or subject's legal representative and ability for study subject to comply with the requirements of the study.
11. Assent from pediatric subjects when appropriate.

Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the integrity of the data.
2. Evidence for more than one seizure focus. (NOTE: For this study, a seizure focus is defined as a cortical region confined to one hemisphere and either one lobe or on a junction of two adjacent lobes from which seizures arise , as documented by scalp or intracranial EEG, that is either supported or not refuted by MRI, and either supported or not refuted by clinical semiology). If the interictal EEG is normal, a seizure focus may be identified by the combination of structural findings on MRI and clinical signs/symptoms associated with the subject's seizures.
3. Seizure focus is one of: interhemispheric, cingulate, or orbitofrontal
4. Seizure focus is hemispheric or poorly defined
5. History of psychogenic nonepileptic seizures in past 2 years, or physiologic nonepileptic seizures and non-epileptogenic events, including suspicion for or a significant history of syncope, and any non-epileptic events must be clearly differentiable from subject's focal seizures based on previously recorded video EEG showing distinct clinical and electrographic features of the subject's PNES compared to their epileptic seizures.
6. Seizures of generalized onset
7. Status epilepticus in the last 12 months
8. Presence of any disease, medical condition or physical condition that, in the opinion of the Investigator, may compromise interfere, limit, affect or reduce the subject's ability to complete a study of 24 weeks duration
9. Presence of any disease, medical condition or physical condition that, in the opinion of the Investigator, may adversely impact the safety of the subject or the integrity of the data.
10. Damaged skin on scalp that may interfere with tDCS stimulation.
11. Pregnant or unwilling to practice birth control during participation in the study.
12. Nursing mothers.
13. Any cranial metal implants (excluding ≦1 mm thick epicranial titanium skull plates and dental fillings) or medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant). Note: Vagus nerve stimulator (VNS) is allowable if the device is in MR Mode (e.g. switched off) during tDCS stimulation and the VNS device is MR conditional.
14. Previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm.
15. A history of addiction to, dependence on, abuse of, misuse of, distribution of, or use of any illicit substance.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The difference between active treatment and sham treatment in the percentage change | from baseline in seizures over the 12 weeks following initiation of treatment.

SECONDARY OUTCOMES:
The proportion of subjects who are responders (defined as subjects with a 50% or greater reduction in seizure frequency | from baseline to week 12 post-treatment

CONTACTS AND LOCATIONS:
Locations (32):
- United States (18):
  - Barrow Neurological Institute, St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Loma Linda University Health, Loma Linda, California
  - Keck Medicine of USC, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of Florida Jacksonville, Jacksonville, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Sinai Hospital, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital Comprehensive Epilepsy Center, Boston, Massachusetts
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Robert Wood Johnson Medical School (Rutgers), New Brunswick, New Jersey
  - University of Rochester, Rochester, New York
  - University of Pennsylvania (Penn Epilepsy), Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, University of Washington, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Ghent University Hospital, Ghent
- France (2):
  - Hospices Civils De Lyon, Lyon
  - CHU de Marseille - Hôpital de la Timone, Marseille
- Spain (10):
  - Hospital Universitario Albacete, Albacete
  - HM Nou Delfos, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Niño Jesús, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Centro de Neurología Avanzada, Seville

IPD SHARING:
Plan to Share IPD: Undecided